CLINICAL TRIAL: NCT05892770
Title: The Effect of Zinc Supplementation Prior to Botulinum Neurotoxin Type A Injection in the Treatment of Spasmodic Dysphonia
Brief Title: Zinc Supplementation Prior to Botox Injections for Spasmodic Dysphonia
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB202202375; OCR43808 (Other: OnCore-UF)
Record Dates: First submitted 2023-04-26; First posted 2023-06-07 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Spasmodic Dysphonia
Keywords: zinc; botox; botulinum toxin; spasmodic dysphonia
MeSH Terms: conditions — Dysphonia | interventions — gluconic acid; Botulinum Toxins, Type A

STUDY DESIGN:
Intervention Model Description: Patient will be followed for one botox cycle as is current standard of care, and another botox cycle with the proposed intervention of zinc supplementation. Each patient will serve as their own control group.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Botulinum toxin A injection (Active Comparator): Botulinum toxin A injection into vocal cords for treatment of spasmodic dysphonia. This is the current standard of care for treatment of this disease process. This will be the control of the study.
  Interventions: Drug: Botulinum toxin type A
- Botulinum toxin A injection +zinc supplementation" (Experimental): Botulinum toxin A injection into vocal cords for treatment of spasmodic dysphonia, with subject taking zinc supplementation daily for the 5 days preceding the botox injection. This will be the experimental arm of the study.
  Interventions: Drug: Zinc gluconate supplement; Drug: Botulinum toxin type A

INTERVENTIONS:
Drug: Zinc gluconate supplement — Subjects will take a 50 mg zinc gluconate supplement at breakfast for the five days leading up to their next injection appointment. They will also answer questionnaires and provide audio recordings at various time points of the two injection cycles, which is roughly six months.
  Other Names: 50 mg zinc gluconate (Puritan's Pride brand)
  Arms: Botulinum toxin A injection +zinc supplementation"
Drug: Botulinum toxin type A — This is the current standard of care for treatment of spasmodic dysphonia. Botox injection goes into the vocal cord muscle, and will be occur in both the control and experimental arms of the study.
  Other Names: Botox Type A

SUMMARY:
One initial study has shown that Botulinum Toxin (BT) in combination with zinc supplementation may increase the duration of effects BT treatment. This initial study was in the context of facial aesthetics. The purpose of the present study is to determine the effect, if any, of oral zinc supplementation prior to BT in the treatment of spasmodic dysphonia. If positive effects will be observed, this would help reduce the burden of disease for these patients.

DETAILED DESCRIPTION:
Botulinum toxin (BT) injections are commonly used to treat various cosmetic, muscular, anesthetic, and neurologic pathologies. In 2012, one study suggested that a combination of zinc and phytase supplementation could increase the duration and degree of effects of botulinum neurotoxin type A (BoNTA). However, this study was met with scientific skepticism due to concerns of financial conflicts of interest, unmasking the study too early, and ambiguity of the dosage of zinc used. In 2021, a new study with 25 patients receiving BoNTA injections for the treatment of excessive gingival display (EGD), showed that zinc supplementation prolonged the effect of BoNTA with statistical significance. There has been no further studies or commentary since these latest results were published. The purpose of this study is to test if the effect of zinc supplementation on BoNTA can be replicated and also translated to a different disease process that is also treated with BT-spasmodic dysphonia (SD). If positive effects are discovered, this would strengthen the preliminary results of the 2021 study, encourage future larger studies on the same hypothesis, and, ultimately, could lead to reducing the burden of disease for patients with SD and any other condition that is treated with BT injections.

ELIGIBILITY:
Inclusion Criteria:

* Adults patients
* 18 years old and above
* Current diagnosis of ADductor spasmodic dysphonia
* Has had Botox injection treatments for SD > 6 months

Exclusion Criteria:

* Pregnant
* Diagnosis of ABductor spasmodic dysphonia
* Patients taking > 30 mg zinc supplementation daily prior to study beginning

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change of Voice-Related Quality of Life (V-RQOL) questionnaire scores during a laryngeal botox injection cycle. | The patient will submit survey on post-injection day 2, 7, 14, 42, 70, and 98. At their next botox injection, a second cycle will immediately begin for an additional 3 months with survey data obtained on post injection day 2, 7, 14, 42, 70, and 98
  10 question, validated questionnaire to assess quality of voice of patients with spasmodic dysphonia. The overall VR-QOL score ranges from 10 to 15 (excellent), 16 to 20 (very good), 21 to 25 (good), 26-30 (fair) and scores more than 30 and up to 50 is poor.
Change in audiometric recording data of subject's speech during a laryngeal botox injection cycle. | The patient record their voice on post-injection day 2, 7, 14, 42, 70, and 98. At their next botox injection, a second cycle will immediately begin for an additional 3 months with audio data obtained on post injection day 2, 7, 14, 42, 70, and 98
  At various points in the study, each subject will be recorded saying the same scripted passage. After all subjects have completed both cycles, all of the accrued audio recordings will be analyzed using a computer algorithm developed by one of our authors that assesses the quality of speech.

CONTACTS AND LOCATIONS:
Overall Officials: Neil Chheda, Principal Investigator — University of Florida
Locations (1):
- University of Florida- Shands Hospital, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No